CLINICAL TRIAL: NCT07012135
Title: Deciphering Preserved Autonomic Function After Multiple Sclerosis
Acronym: DPAF-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan J. Solinsky, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-007459
Record Dates: First submitted 2025-05-14; First posted 2025-06-10 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Control Subjects; Autonomic Dysreflexia
MeSH Terms: conditions — Multiple Sclerosis; Autonomic Dysreflexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with multiple sclerosis (Experimental)
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of sympathetic activation; Diagnostic Test: Testing of autonomic dysreflexia
- Individuals without multiple sclerosis (Experimental)
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of sympathetic activation; Diagnostic Test: Testing of autonomic dysreflexia

INTERVENTIONS:
Diagnostic Test: Tests of sympathetic inhibition — Bolus phenylephrine infusion using the Oxford technique will generate the need to inhibit sympathetic activity. Similarly, resting state Mayer waves will be assessed with regard to heart rate and blood pressure responses.
Diagnostic Test: Tests of sympathetic activation — Cold pressor test of the hand will be used to cause sympathetic activation. Valsalva's maneuver will assess the ability to buffer against blood pressure fall (phase II).
Diagnostic Test: Testing of autonomic dysreflexia — Cold pressor test of the foot and bladder pressor response will be tested.

SUMMARY:
This study looks to characterize gradients of dysfunction in the autonomic nervous system in patients with clinically diagnosed multiple sclerosis. The autonomic nervous system plays key roles in regulation of blood pressure, skin blood flow, and bladder health- all issues that individuals with multiple sclerosis typically suffer. Focusing on blood pressure regulation, the most precise metric with broad clinical applicability, the investigators will perform laboratory-based tests to probe the body's ability to generate autonomic responses. For both individuals with multiple sclerosis and uninjured controls, laboratory-based experiments will utilize multiple parallel recordings to identify how the autonomic nervous system is able to inhibit and activate signals. The investigators anticipate that those with autonomic dysfunction with multiple sclerosis will exhibit abnormalities in these precise metrics. The investigators will look to see if any substantial connections exist between different degrees of preserved autonomic function and secondary autonomic complications from multiple sclerosis. In accomplishing this, the investigators hope to give scientists important insights to how the autonomic nervous system works after multiple sclerosis and give physicians better tools to manage these secondary autonomic complications.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* clinically confirmed diagnosis of multiple sclerosis -OR- uninjured control

Exclusion Criteria:

* symptoms of cardiovascular (including, but not limited to: hypertension, stroke, chest pain, etc.), respiratory, peripheral neurological or autonomic disease (particularly diabetes mellitus requiring treatment)
* women who are pregnant or lactating
* having a body mass index (BMI) ≥ 35 kg/m2
* taking or being administered a medication known to potentially have adverse interactions with phenylephrine
* in the judgement of the principal investigator or clinical collaborator, any illness or condition that will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Valsalva Maneuver Phase II | During single laboratory diagnostic testing session, on average 30 minutes after start of laboratory testing session
  Presence or absence of phase II on Valsalva maneuver testing, which takes approximately 15 seconds to complete. This will be repeated x3.

SECONDARY OUTCOMES:
Beat-to-beat heart rate | Continuous recording during single laboratory diagnostic testing session, from baseline to lab session end, average of 3 hours in duration
  Electrocardiogram will record continuous measures with changes in R-R interval (ms) quantified and compared to baseline.
Beat-to-beat blood pressure | Continuous recording during single laboratory diagnostic testing session, from baseline to lab session end, average of 3 hours in duration
  Non-invasive continuous blood pressure monitors will be used, with changes in systolic and diastolic pressure (in mmHg) from resting baseline measured.
Quantify autonomic dysreflexia and orthostatic hypotension | Baseline, prior to laboratory diagnostic testing session
  Participants will be given the Autonomic Dysfunction Following Spinal Cord Injury questionnaire (score range 0-436, with higher scores indicating more autonomic dysfunction).
Quantify secondary autonomic complications | Baseline, prior to laboratory diagnostic testing session
  Participants will be given the Composite Autonomic Symptom Score (range 0-100, with higher scores indicating more autonomic dysfunction).
Serum Catecholamines | 3x during single laboratory diagnostic testing session - collected at Baseline, pre-pressor test, post-pressor test - pre-pressor & post-pressor timepoint labs collected on average 2.5 & 3 hours post-baseline, respectively
  A series of 3 serum catecholamine draws will occur during the study visit at baseline, pre-pressor test, and post-pressor test to evaluate change in stress hormone.
Serum Cortisol | 3x during single laboratory diagnostic testing session - collected at Baseline, pre-pressor test, post-pressor test - pre-pressor & post-pressor timepoint labs collected on average 2.5 & 3 hours post-baseline, respectively
  A series of 3 serum cortisol draws will occur during the study visit at baseline, pre-pressor test, and post-pressor test to evaluate change in stress hormone.
T-Cell Exhaustion Markers | During single laboratory diagnostic testing session - Baseline
  Blood will be drawn at start of laboratory testing to assess T-cell exhaustion markers by incidence of surface markers including PD-1, TIM-3, LAG3, and CTLA-4 per individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No